CLINICAL TRIAL: NCT01402739
Title: Monocentric Pilot Study of Algorithm-Guided Transfusions in Cardiac Surgery Patients for Reduction of Drainage Blood Losses
Brief Title: Algorithm-Guided Transfusions in Cardiac Surgery Patients for Reduction of Drainage Blood Losses
Acronym: HEART-PoC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated prematurely due to futility
Sponsor: Michael Sander (Other)
Responsible Party: Sponsor-Investigator, Michael Sander, Univ.-Prof. M. Sander, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEART-PoC
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Chest Tube Output; Allogeneic Blood Transfusions
Keywords: PoC; ROTEM; Multiplate; transfusion; cardiac surgery; drainage blood loss; chest tube output

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PoC algorithm guided transfusions (Experimental): experimental arm
  Interventions: Other: Point of Care Coagulation Monitoring Guided Transfusion Algorithm
- standard of care transfusions (Active Comparator): control arm
  Interventions: Other: standard coagulation monitoring guided transfusion algorithm

INTERVENTIONS:
Other: Point of Care Coagulation Monitoring Guided Transfusion Algorithm — (thromboelastometry, aggregometry, blood gas analysis)
  Other Names: ROTEM delta, Multiplate, ABL 725
  Arms: PoC algorithm guided transfusions
Other: standard coagulation monitoring guided transfusion algorithm — aPTT, ACT, platelet count, hemoglobin, fibrinogen
  Arms: standard of care transfusions

SUMMARY:
Cardiac surgery patients have a risk to need allogeneic blood transfusions that depends on several risk factors, e.g. the type of surgery, concomitant medication with anticoagulants, and postoperative chest tube output. Allogeneic blood transfusion is associated with transfusion reactions, infection transmission, and postoperative morbidity and mortality. The aim of this study is to investigate, whether cardiac surgery patients have a reduced postoperative chest tube output and transfusion need when using a point-of-care guided transfusion algorithm compared to standard of care transfusion protocols.

DETAILED DESCRIPTION:
Cardiac surgery patients have a risk to need allogeneic blood transfusions that depends on several risk factors, e.g. the type of surgery, concomitant medication with anticoagulants, and postoperative chest tube output. Allogeneic blood transfusion is associated with transfusion reactions, infection transmission, and postoperative morbidity and mortality. The aim of this study is to investigate, whether cardiac surgery patients have a reduced postoperative chest tube output and transfusion need when using a point-of-care guided transfusion algorithm compared to standard of care transfusion protocols .

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery patient requiring cardiopulmonary bypass
* moderate or high transfusion risk
* signed informed consent

Exclusion Criteria:

* age <18 or >80 years
* known hemophilia
* known thrombophilia
* known thrombocytopathy
* hereditary or acquired coagulation disorder
* active endocarditis
* ejection fraction <30%
* BSA < 1.8 sqm
* planned aortic arch surgery
* preoperative thrombocytopenia <150/nl
* underlying hemostaseological disease
* preoperative anemia
* liver cirrhosis Child B or higher
* preoperative creatinine > 2mg/dl
* terminal renal insufficiency requiring dialysis
* vitamin k antagonists during 5 days prior to surgery
* pregnant or breast-feeding women
* known allergy against allogeneic blood products or coagulation factors
* refusal of blood transfusions
* any concomitant investigational agent or participation in another trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
chest tube output | 24 hours

SECONDARY OUTCOMES:
need of allogeneic blood transfusions | 24 hours
course of conventional coagulation parameters (aPTT, TPZ, fibrinogen, FXIII, ACT) | 24 hours
duration of mechanical ventilation | hours (average)
incidence of RRT | during 30 days
  or until hospital discharge, whatever is earlier

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sander, MD, Principal Investigator — Dept. of Anesthesiology CCM/CVK Charité Universitätsmedizin Berlin; Claudia D Spies, MD, Study Chair — Dept. of Anesthesiology CCM/CVK Charité Universitätsmedizin Berlin
Locations (1):
- Department of Anesthesiology CCM/CVK Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Lehmann F, Rau J, Malcolm B, Sander M, von Heymann C, Moormann T, Geyer T, Balzer F, Wernecke KD, Kaufner L. Why does a point of care guided transfusion algorithm not improve blood loss and transfusion practice in patients undergoing high-risk cardiac surgery? A prospective randomized controlled pilot study. BMC Anesthesiol. 2019 Feb 18;19(1):24. doi: 10.1186/s12871-019-0689-7. PMID 30777015